CLINICAL TRIAL: NCT01433887
Title: Response to Pegylated Interferon and Ribavirin in Chinese Patients With Chronic
Brief Title: Response to Pegylated Interferon and Ribavirin in Chinese Patients With Chronic Hepatitis C Genotypes 1 Versus 2/3 Versus 6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Cai Qingxian, Sun Yat-Sen University, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAH5010G6HCV
Record Dates: First submitted 2011-09-11; First posted 2011-09-14 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Hepatitis C
Keywords: Peginterferon alfa-2a; ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Genotype 6 (Experimental): Genotype 6 chronic hepatitis C patients will be treated with Peginterferon alfa-2a plus ribavirin for 48 weeks
  Interventions: Drug: 48-weeks course; Drug: Ribavirin
- Genotype 1 (Experimental): Genotype 1 chronic hepatitis C patients will be treated with Peginterferon alfa-2a plus ribavirin for 48 weeks
  Interventions: Drug: 48-weeks course; Drug: Ribavirin
- Genotype 2/3 (Experimental): Genotype 2/3 chronic hepatitis C patients will be treated with Peginterferon alfa-2a/2b plus ribavirin for 24 weeks
  Interventions: Drug: Peginterferon alfa2a; Drug: Ribavirin

INTERVENTIONS:
Drug: 48-weeks course — patients receive a dose of 180 µg of PEGASYS once a week for 48 weeks
  Arms: Genotype 1; Genotype 6
Drug: Ribavirin — patients receive a dose 800 to 1200 mg of ribavirin once a day(according to weight) for 48 weeks
  Arms: Genotype 1; Genotype 6
Drug: Peginterferon alfa2a — patients receive a dose of 180 µg of PEGASYS once a week for 24 weeks
  Arms: Genotype 2/3
Drug: Ribavirin — patients receive a dose 800 to 1200 mg of ribavirin once a day(according to weight) for 24 weeks
  Arms: Genotype 2/3

SUMMARY:
The Chinese patients with chronic hepatitis C have a different genetic background, which had been demonstrated to significantly influence their responses to pegylated interferon and ribavirin. In this study, Chinese patients with Hepatitis C Virus genotype 1, 2/3, 6 infection were treated with pegylated interferon and ribavirin. Their response was compared amongst different genotypes.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA is positive
* Treatment naive
* Come from China

Exclusion Criteria:

* Active substance abuse
* Poorly controlled psychiatric disease
* HBsAg positive
* Anti-HIV positive
* Suffering from other significant concurrent medical conditions including chronic liver diseases

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) | 24 weeks after the end of treatment
  Undetectable HCVRNA in serum(<15IU/ml) 24 weeks after the end of treatment

SECONDARY OUTCOMES:
Change in health related quality as measured by short form 36 (SF-36) from baseline to 24 weeks after the end of treatment | 24 weeks after the end of treatment
Sick leave in patients treated for 24 or 48 weeks treatment | 48 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Eighth People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Zhongshan second people's hospital, Zhongshan, Guangdong